CLINICAL TRIAL: NCT03408964
Title: An Exploratory proof-of Valid Biomarkers in Blood to Predict the Response to Therapy in Prostate Cancer Patients, a Single Center Study
Brief Title: Valid Biomarkers in Blood to Predict the Response to Therapy in Prostate Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor
Other Study IDs: IOSI-IOR-002
Record Dates: First submitted 2018-01-11; First posted 2018-01-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Group 0 (set-up): Patients with known diagnosis of CSPC (Group 0a) and CRPC (Group 0b) irrespective of the PC treatment (not first diagnosis)
  Interventions: Other: biological samples collection and analysis
- Group 1a (control): Patients who underwent biopsies for suspected Prostate Cancer (PC), with a negative result for invasive cancer
  Interventions: Other: biological samples collection and analysis
- Group 1: Patients with a first diagnosis of localized biopsy-proven PC, untreated, planned to undergo radical surgery and / or radical radiotherapy
  Interventions: Other: biological samples collection and analysis
- Group 2: Patients with a diagnosis of locally advanced unresectable, recurrent or metastatic PC planned to receive first-line hormono therapy
  Interventions: Other: biological samples collection and analysis
- Group 3: Patients with recurrent/progressive/metastatic CRPC planned to receive chemotherapy
  Interventions: Other: biological samples collection and analysis
- Group Exo: Patients with a known or suspected diagnosis of PC or at any stage of the disease and irrespective of the treatment undergoing an imaging investigation.
  Interventions: Other: biological samples collection and analysis
- Group Bio: Patients with a known or suspected diagnosis of PC at any stage of the disease and irrespective of the treatment undergoing a tumour sampling.
  Interventions: Other: biological samples collection and analysis

INTERVENTIONS:
Other: biological samples collection and analysis — Participants to the study will be assigned to 4 cohorts according to the stage of disease and planned antitumor treatment at time of study entry; they will be followed up and sampled according to a defined time schedule

SUMMARY:
Participants to the study will be assigned to 7 cohorts according to the stage of disease and planned antitumor treatment at time of study entry.

In all patients, 12 ml of blood sample will be collected in EDTA tube for analysis of biological biomarkers in different time points.

DETAILED DESCRIPTION:
Participants to the study will be assigned to 5 cohorts according to the stage of disease and planned antitumor treatment at time of study entry.

Group 0 (set-up): blood sampling and rectal swab will be collected at a single time-point during the PC treatment. No follow-up is required.

Group 1a (control): the first blood sampling will be performed within 4 weeks since the negative biopsy; subsequent samplings will be done according to a schedule comparable to that of Group 1 up to 1 year or evidence of tumor, whichever occurs first.

Group 1, Group 2 and Group 3: the first blood sampling will be performed before radical treatment or HT start or CT start, on the basis of the planned antitumor therapy; subsequent sampling will be done after radical intervention at 4 weeks (only for Group 1) and then every 3 months (or more frequently if clinically indicated), up to 3 years or evidence of tumor recurrence/progression (radiological or biochemical), whichever occurs first.

At the time of recurrence/progression, patients of Group 1 could become part and could be followed as per Group 2, and patients of Group 2 could become part and could be followed as per Group 3.

Group Exo and Group Bio: blood sampling will be performed at a single time-point during the PC treatment. No follow-up is required.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria (for entering all groups)

* Age ≥ 18 years
* Histological diagnosis of prostate adenocarcinoma at different stages of disease (see Section 6.2) for which a treatment is indicated
* Written Informed Consent

Inclusion criterion only for entering Group 0

• Patients with a known diagnosis of CSPC or CRPC

Inclusion criterion only for entering Group 1a

• Patients that underwent biopsies for a suspect of PC, but resulted negative for cancer

Exclusion Criteria:

General exclusion criteria (for entering all groups)

* Active infection requiring treatment
* Decrease of general condition
* Concomitant severe comorbities
* Difficult socioeconomic conditions making regular follow up unfeasible.
* Need of concomitant steroids at study entry and during the study
* Diagnosis of second tumor in the previous 5 years

Exclusion criterion only for entering Group 0

• No antibiotic treatments in the previous 2 months before enrollment

Exclusion criteria only for entering Group 1

* Previous radical surgery and / or radical radiotherapy
* Previous hormonal treatments

Exclusion criteria only for entering Group 2

* No antibiotic treatments in the previous 2 months before enrollment (only in patients enrolling also for metagenomics and metabolomics)
* Previous hormonal treatments for advanced disease

Exclusion criterion only for entering Group 3

• No antibiotic treatments in the previous 2 months before enrollment (only in patients enrolling also for metagenomics and metabolomics analyses)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate adenocarcinoma at different stages of disease
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers value in the response to therapy | 3 years
  To assess the value of MDSCs, NLR, cytokines as biomarkers of clinical outcome at different stages of disease and their correlation with PSA, the marker usually used for PC

SECONDARY OUTCOMES:
Biomarkers inter and intra variability | 3 years
  to assess the inter- and intra-variability of the value of MDSCs, NLR and cytochines.
Metabolomic and metagenomic analysis | 3 years
  to set-up the microbiota analysis and blood analysis quantification and determine the intra- and inter-patient variability (Group 0);
Metabolomic and metagenomic analysis | 3 years
  to assess the diversity and the composition of the intestinal microbiota and its blood metabolites in PC patients in castration-sensitive (Group 2) and castration-resistant (Group 3) phase

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Pereira Mestre, MD, Principal Investigator — Oncology Institute of Southern Switzerland (IOSI)
Locations (1):
- Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Switzerland